CLINICAL TRIAL: NCT05521737
Title: Effect of Electroacupuncture on Sensitive Symptoms of Distal Diabetic Peripheral Neuropathy and Its Correlation With Nerve Conduction Changes
Brief Title: Effect of Electroacupuncture on Sensitive Symptoms of Distal Diabetic Peripheral Neuropathy
Acronym: EA&DPN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: National Polytechnic Institute, Mexico (Other); Instituto Nacional de Salud Publica, Mexico (Other); Escuela Superior de Medicina, Instituto Politécnico Nacional (Unknown); Escuela Nacional de Medicina y Homeopatía, Instituto Politécnico Nacional (Unknown); Universidad Nacional Autonoma de Mexico (Other); Facultad de Estudios Superiores Iztacala, Universidad Nacional Autónoma de Mexico (Unknown); Facultad de Estudios Superiores Zaragoza, Universidad Nacional Autónoma de Mexico (Unknown); Facultad de Medicina, UNAM (Unknown)
Responsible Party: Principal Investigator, José de Jesús Peralta Romero, Principal investigator, head of clinical department of the Medical Research Unit in Biochemistry, UMAE, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-2020-785-070; 09-CEI-009-20160601 (Other: CONBIOÉTICA); 17 CI 09 015 006 (Other: COFEPRIS)
Record Dates: First submitted 2022-08-22; First posted 2022-08-30 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Electroacupuncture; Acupuncture; Diabetic Polyneuropathy; Diabetic Peripheral Neuropathy; Diabetic Peripheral Neuropathic Pain; Nerve Conduction
Keywords: Electroacupuncture; Acupuncture; Diabetic Polyneuropathy; Diabetic Peripheral Neuropathy; Diabetic Peripheral Neuropathic Pain; Nerve Conduction; Diabetic Pain
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Electroacupuncture; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: The protocol consists of two study groups, including a control group of sham acupuncture, and an interventional group of Electroacupuncture. Both interventions will be applied in a total of 32 sessions, divided into two intervention cycles, that is, 16 sessions over two months, with a rest period of one month in between. ,Acupuncture points are Zusanli (E36), Fenlong (E40), Yinlingquan (B9), Sanyinjiao (B6), Taichong (H3) and Zulinqi (VB41).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patient masking: During the application of the intervention, a bandage is placed over the patients eyes so that the participants cannot see the type of therapy applied (electroacupuncture or sham acupuncture).
  Statistical masking: The researcher in charge of the statistical analysis is unaware of the type of intervention received by the patients and delivers the results to the responsible researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham group (Sham Comparator): Sham acupuncture will be administered in a total of 32 sessions within five months.
  Interventions: Procedure: Sham Acupuncture
- Interventional group (Experimental): Electroacupuncture will be administered in a total of 32 sessions within five months.
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — Intervention consists of a total of 32 sessions, divided into two intervention cycles, that is, 16 sessions over two months, with a rest period of one month in between. EA is applied for 20 minutes at an alternating frequency of 2 Hz. Acupunctural points are Zusanli (E36), Fenlong (E40), Yinlingquan (B9), Sanyinjiao (B6), Taichong (H3) and Zulinqi (VB41).
  Other Names: EA
  Arms: Interventional group
Procedure: Sham Acupuncture — Intervention consists of a total of 32 sessions, divided into two intervention cycles, that is, 16 sessions over two months, with a rest period of one month in between. Sham acupuncture will be applied using a nonpuncture device without electrical stimulation at the same acupunctural points as in the EA group.
  Other Names: Sham
  Arms: Sham group

SUMMARY:
This is a controlled clinical trial with the aim to study the effects of electroacupuncture on neuropathic pain reduction, quality of life and changes in sensory and motor nerve conduction velocity in patients with type 2 diabetes mellitus, beneficiaries of the familiar medical centers 20, 40 and 41 of the Instituto Mexicano del Seguro Social, at north of Mexico City, in colaboration with the human acupuncture specialty of the Escuela Nacional de Medicina y Homeopatía, Instituto Politécnico Nacional, Mexico.

DETAILED DESCRIPTION:
Controlled clinical trial to evaluate the effect of electroacupuncture on the reduction of neuropathic pain, quality of life; electrophysiological, inflammatory response, oxidative stress, and genetic expression, in patients with type 2 diabetes mellitus, beneficiaries from the family medical centers 20 , 40 and 41 of the Instituto Mexicano del Seguro Social, at north of Mexico City.

Once the acceptance letter has been signed, a series of questionnaires (MNSI, MDNS, DN-4, NRS, and SF-36), and a physical examination will be carried out to meet the necessary criteria to continue participating.

Only candidates with clinical diagnosis of diabetic polyneuropathy will have an electrophysiological examination by nerve conduction velocity study, if so, patients will be randomized to the electroacupunture or sham acupuncture groups.

Before intervention, laboratory studies will be taken after fasting for 8 to 10 hours, to determine biochemichal profile (glucose, urea, creatinine, uric acid , triglycerides, total cholesterol, HDL and LDL), oxidative stress (Malondialdehyde), inflammatory response (IL-6, IL1β, TNF-α, IL-10 and IL-18 cytokines), and gene expression (5-HT1AR, Neurokinin 1, α-adrenoreceptors, NGF, CX3CR1, GAP-43, and NT3).

Intervention will be applied in a total of 32 acupuncture sessions, divided into two intervention cycles, that is, 16 sessions over two months, with a rest period of one month in between.

At the end of both cycles of interventions, the questionnaires, the nerve conduction velocity study the biochemical and molecular studies will be re-assessed. Finally, this will be re-evaluated after three months post-intervention in order to evaluate the effect of intervention over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes.
* Patients with clinical diabetic peripheral polyneuropathy.
* Patients with electrophysiological diagnosis of diabetic peripheral polyneuropathy in its different types of classification.

Exclusion Criteria:

* Type 1 Diabetes or gestational diabetes.
* Systemic autoimmune diseases.
* Hematological disorders.
* HIV diagnosis.
* Cancer in treatment.
* Pregnancy.
* Other types of neurological disorders or neuropathies.
* Intervention with acupuncture six months previously.
* Patients with pacemarkers.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Nerve Conduction Velocity | Baseline evaluation, after the first and second cycle of intervention, respectively, and three months after the end of the intervention.
  Measured by Nerve Conduction Velocity Study using the VIKING LIFE-SAVING EQUIPMENT, to determine Motor and Sensitive Nerve Conduction Velocity of common peroneal nerve, sural nerve, and tibial nerve.
  Sensitive Nerve Conduction (SCV). Distance between the receiving point and the stimulus point. SCV normal values: Peroneal nerve ≥ 41 m/s, tibial nerve ≥ 44 m/s, sural nerve ≥ 50 m/s.
  Motor Conduction Velocity (MCV). Distance between two points and the difference in incubation between them after superstimulation of the corresponding nerve branch. MCV normal values: Peroneal nerve ≥ 41 m/s, tibial nerve ≥ 44 m/s, sural nerve ≥ 60 m/s.
  *Values below those stipulated above indicate that NCV has slowed down, and is abnomal.
  The investigators expect a diminishment of SCV and MCV in sham acupuncture group from the first cycle of intervention whereas electroacupuncture group remains unchanged or even increases SCV and MCV.

SECONDARY OUTCOMES:
Michigan Neuropathy Screening Instrument (MNSI). | Baseline evaluation, after the first and second cycle of intervention, respectively, and three months after the end of the intervention.
  It will be assessed with a lower extremity examination by a health professional of both feet in search of deformities, dry skin, calluses, infections, fissures and ulcers. Complemented with measurement of vibratory sensation, ankle reflexes, and Semmes-Weinstein monofilament test.
  The investigators expect improvement in the physical aspect of the foot in the electroacupuncture group, while in the sham acupuncture group the complication progresses.
Michigan Diabetic Neuropathy Score (MDNS) | Baseline evaluation, after the first and second cycle of intervention, respectively, and three months after the end of the intervention.
  Composed of three items where the sensory compromise is evaluated with the perception of vibration, 10 gr. monofilament and pin prick, in addition to the muscular strength of the toes, and the bicipital, tricipital, quadriceps and achilles muscle reflexes. The investigators expect a diminishment of MDNS score and clinical improvement in the electroacupuncture group and progression of clinical manifestations in the sham group.
Douleur Neuropathique en 4 Questions (DN-4) | Baseline evaluation, after the first and second cycle of intervention, respectively, and three months after the end of the intervention.
  A screening tool for neuropathic pain consisting of 10 interview questions (DN4-interview) and physical tests. A score greater than 4 points suggests neuropathic pain. The investigators expect decreased scores in the electroacupuncture group and increased or persistent scores in the sham group.
Numerical Pain Rating Scale (NRS) | Baseline evaluation, after the first and second cycle of intervention, respectively, and three months after the end of the intervention.
  Patients are only asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that best matches the intensity of their pain currently and in the last 7 days, where zero usually represents "no pain", while the upper limit represents "the worst pain of their life". The investigators expect diminishment of rating scale in electroacupuncture group and an increase in sham acupuncture group.
Quality life (SF-36) | Baseline evaluation, after the first and second cycle of intervention, respectively, and three months after the end of the intervention.
  It will be measured by The Short Form-36 Health Survey (SF-36) a measure of health status that consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health), which are the weighted sums of the questions in their section. The investigators expect quality life improvement in electroacupuncture group while in sham acupuncture group might worsen.
Oxidative Stress | Baseline evaluation, after the first and second cycle of intervention, respectively, and three months after the end of the intervention.
  Determined by quantifying the concentrations of the lipoperoxidation product Malondialdehyde (MDA). An increase of MDA is expected in the sham group, while in the electroacupuncture group it is expected to decrease.
Inflammatory response | Baseline evaluation, after the first and second cycle of intervention, respectively, and three months after the end of the intervention.
  Assessed by changes in serum concentrations of proinflammatory (IL-6, IL1β, TNF-α and IL-18) and anti-inflammatory (IL-10) cytokines determined by quantitative ELISA by flow cytometry. The investigators expect increase of anti-inflammatory cytokine and decrease of proinflammatory cytokines in the electroacupuncture group, while in the sham group this is inversely presented.
Genetic expression | Baseline evaluation, after the first and second cycle of intervention, respectively, and three months after the end of the intervention.
  mRNA expression of 5-HT1AR, Neurokinin 1, α-adrenoreceptors, NGF (Nerve growth factor), CX3CR1, GAP-43 (Growth associated protein 43) and Neurotrophin (NT3), (Chemoline receptor 1) genes quantified by real-time PCR. The investigators expect an increase in gene expression in patients with electroacupuncture while in sham patients it is decreased or even unchanged.

CONTACTS AND LOCATIONS:
Overall Officials: José de Jesús Peralta Romero, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Medical research unit in biochemistry, UMAE "Dr. Bernardo Sepúlveda".Centro Médico Nacional Siglo XXI, Instituto Mexicano del Seguro Social., Mexico City, Cuauhtémoc, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez Hernandez MF, Calderon Vallejo A, Aguilar Castillo SJ, Gomez Jimenez DC, Rodriguez Guerrero E, Aguilar Morales F, Moreno Tovar MG, Zurita Munoz MA, Bautista Cortez AE, Calzada Mendoza CC, De Nova Ocampo MA, Ordonez Rodriguez JM, Gomez Esquivel ML, Garcia Mendez A, Flores Gil O, Macias Zaragoza VM, Cortes Moreno GY, Salinas Lara C, Velazquez Garcia G, Saldivar Ceron HI, Perez Navarro LM, Avila Jimenez L, Gomez Zamudio JH, Diaz Flores M, Cruz Lopez M, Ocharan Hernandez ME, Peralta Romero JJ. Electroacupuncture efficacy in diabetic polyneuropathy: Study protocol for a double-blinded randomized controlled multicenter clinical trial. BMC Complement Med Ther. 2024 Feb 15;24(1):90. doi: 10.1186/s12906-024-04375-8. PMID 38360684
- [Derived] Perez Hernandez MF, Rodriguez Guerrero E, Ocharan Hernandez ME, Gomez Jimenez DC, Gomez Esquivel ML, Aguilar Castillo SJ, Flores Hernandez VD, Romo Duenas S, Torres Mendoza MR, Calderon Vallejo A, Velazquez Garcia G, Moreno Tovar MG, Cruz Lopez M, Ordonez Rodriguez JM, Pena Juarez KA, Miranda Gastelum X, Castro Diaz JM, Aguirre Guerrero A, Macias Zaragoza VM, Peralta Romero JJ. Effect of electroacupuncture for pain relief in diabetic distal symmetric polyneuropathy: a pilot randomized clinical trial. BMC Complement Med Ther. 2025 Dec 9;25(1):438. doi: 10.1186/s12906-025-05135-y. PMID 41366387
- Available data/document: Protocol reapproval report — https://drive.google.com/file/d/1P3sbgleW3murWJq_FIaerBlFU12aga9z/view?usp=sharing

DOCUMENTS (7):
  • Study Protocol: COMITEE PROTOCOL REAPPROVAL 2022 - 2023 (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT05521737/Prot_000.pdf
  • Study Protocol: COMITEE PROTOCOL APPROVAL 2020 - 2021 (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT05521737/Prot_001.pdf
  • Study Protocol: COMITEE PROTOCOL REAPPROVAL 2021 - 2022 (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT05521737/Prot_002.pdf
  • Study Protocol: Publication of Study Protocol (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT05521737/Prot_005.pdf
  • Study Protocol: RESEARCH COMITEE PROTOCOL REAPPROVAL 2023 - 2024 (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT05521737/Prot_006.pdf
  • Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT05521737/SAP_003.pdf
  • Informed Consent Form (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT05521737/ICF_004.pdf